CLINICAL TRIAL: NCT05337423
Title: Photobiomodulation in the Treatment of Palmar-plantar Erythrodysesthesia: Clinical, Randomized, Controlled Study
Brief Title: Photobiomodulation in the Treatment of Hand-foot Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment over one year resulted in only six patients treated. With the conclusion of the principal investigator's doctoral program and limited resources to continue, the study was terminated due to time and availability constraints.
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UninoveUCU
Record Dates: First submitted 2022-04-04; First posted 2022-04-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Erythrodysesthesia Syndrome
Keywords: Hand-Food Syndrome; Low-Level Light Therapy; Quality of life
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: A Group of participants will receive skin moisturizer and photobiomodulation sham while another group will receive the skin moisturizer and the active photobiomodulation treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participants involved in the study, nor the outcomes assessor will be aware of the groups formed, as well as the treatments received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Moisturizing cream indicated and provided by the hospital (with urea) + LED treatment.
  Interventions: Device: Photobiomodulation; Other: Moisturizer
- Group 2 (Sham Comparator): Moisturizing cream indicated and provided by the hospital (with urea) + LED sham treatment.
  Interventions: Other: Moisturizer

INTERVENTIONS:
Device: Photobiomodulation — Group 1 will receive 630 nm LED and group 2 will receive sham treatment twice a week in the palmo-plantar areas of the hands and feet (4 J/cm2) for 4 weeks.
  Other Names: low-level laser therapy
  Arms: Group 1
Other: Moisturizer — Both groups will receive moisturizer.

SUMMARY:
A cytotoxic complication caused by chemotherapy is hand-foot syndrome, also known as palmar-plantar erythrodysesthesia (PPE). The mechanism is not yet clear, but it is thought that the chemotherapeutic agent generates cytotoxicity on the acral epidermis. Clinically it manifests as erythema and edema on the palms of the hands and feet, dry and scaly skin, accompanied by a sensation of tightness and pain. Extreme cases present blisters and ulcerations that may require hospitalization. It can also be accompanied by paresthesias. The main objective will be to evaluate if photobiomodulation is effective in reducing PPE induced by Capecitabine and 5-Fluorouracil chemotherapy.

It will be a 4 week treatment, with 2 groups: G1 - Moisturizing cream and Photobiomodulation; G2: Moisturizing cream and photobiomodulation sham.

DETAILED DESCRIPTION:
Methodology: randomized, controlled, double-blind, single-center clinical trial. The study population (40 participants) will be divided into two groups - Group 1: moisturizer plus LED (light emitting diode) treatment and Group 2: moisturizer plus LED sham treatment. For the application of LED light, Antares (ibramed) with P2 LED cluster (630 nm) will be applied twice a week in the palmo-plantar areas of the hands and feet (4 J/cm2) for 4 weeks.

The Palmar-plantar Erythrodysesthesia (PPE) degree is the main outcome while the secondary outcomes are the data referring to the chemotherapy treatment plan (Chemotherapy dose, need of reducing drug dose or interrupting the treatment) and also the quality of life by using Hand-foot syndrome (HSF) questionnaire - HSF-14 and dermatology Life Questionnaire Index (DLQI). PPE grade and chemotherapy plan will be measured prior to the start of treatment with photobiomodulation, in the middle and at the end of it. Quality of life questionnaires (HFS-14 - Hand-foot syndrome and DLQI - dermatology Life Questionnaire Index) will be applied at the beginning and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* hospitalized or outpatients,
* with oncological pathology (confirmed by anatomo-pathological or cytological diagnosis)
* undergoing chemotherapy treatment (oral capecitabine and 5-Fluorouracil in continuous infusion, following the treatment plans protocolized by the institution: Xelox Bevacizumab, Capecitabine, Capecitabine + Radiotherapy, Folfoxiri, Xeliri-Bevacizumab, Folfox4-Bevacizumab , Docetaxel-CDDP-5-Fluorouracil (Colony Stimulating Factors), mFolfirinox q/14 days, Flot.)
* who develop hand-foot syndrome of greater or equal toxicity to 1 on the CTC scale NCI v. 5.0 and on Saif scale. Et al. for dark skin

Exclusion Criteria:

* Patients with palmo-plantar skin comorbidities,
* autoimmune comorbidities,
* amputated limbs,
* systemic infection,
* localized or regional limb infection,
* respiratory isolation,
* contact isolation
* insulin-requiring diabetics.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Palmo planar erythrodysesthesia grade | Before treatment (Day 0), at half treatment (Day 14) and at the end of the treatment (Day 28)
  3 Epp grades were stablished by CTC NCI being: Grade 1 - Minimal palmoplantar skin changes, without pain (erythema, edema, hyperkeratosis),; grade 2 - Skin changes (scaling, blisters, fissures, edema, hyperkeratosis) with pain, limiting instrumental activities; grade 3 - Severe skin changes (scaling, blisters, fissures, edema, hyperkeratosis, bleeding), with pain..

SECONDARY OUTCOMES:
Chemotherapy dose | Before treatment (Day 0), at half treatment (Day 14) and at the end of the treatment (Day 28)
  Total dose (mg) of chemotherapeutical drug used
Need of interrupting chemotherapy | Before treatment (Day 0), at half treatment (Day 14) and at the end of the treatment (Day 28)
  The need of interrupting chemotherapy due to Palmo planar erythrodysesthesia : Yes or no
Need of reducting chemotherapy dose | Before treatment (Day 0), at half treatment (Day 14) and at the end of the treatment (Day 28)
  The need of reducing dose of chemotherapy due to Palmo planar erythrodysesthesia: Yes or no
HSF-14 | Before treatment (Day 0) and at the end of the treatment (Day 28)
  Quality of life questionnaire HSF-14
DLQI | Before treatment ( Day 0) and the end of the treatment (Day 28)
  Quality of life questionnaire - Dermatology life quality index
Questionnaire | Follow up (day 60)
  Questionnaire developed by researchers evaluating parameters in hands and feet related to daily activities.
Peripheral Sensory Neuropathy World Health Organization (WHO) Scale | Before treatment ( Day 0) and the end of the treatment (Day 28)
  Peripheral Sensory Neuropathy World Health Organization (WHO) Scale Grade 0: No; grade 1: symptoms Presence of paresthesias and/ or decreased deep tendon reflexes; Grade 2: Severe paresthesias and/or light muscle weakness Grade 3: Intolerable paresthesias and/or marked weakness , Grade 4: Paralysis
Peripheral Sensory Neuropathy Eastern Clinical Oncology Group (ECOG) Scale | Before treatment ( Day 0) and the end of the treatment (Day 28)
  Peripheral Sensory Neuropathy Eastern Clinical Oncology Group (ECOG) Scale Grade 0, None, or no change; Grade 1: Loss of deep tendon reflexes, mild paresthesias. Grade 2: Mild or moderate objective sensory loss; moderate paresthesias. Grade 3: Severe objective sensory loss, or paresthesias that interfere with function

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Lestido, Master, Principal Investigator — Universidad Catolica de Uruguay
Locations (2):
- Uruguay (2):
  - Centro de Asistencia del Sindicato Médico del Uruguay, Montevideo
  - Instituto Nacional del Cáncer, Montevideo

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared. The sharing will begin 3 months following article publication. Researchers who provide a methodologically sound proposal will receive the access. Proposals should be directed to chrispavani@gmail.com. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.Proposals should be directed to xxx@yyy. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Derived] Lestido V, Rodriguez F, Rodriguez A, Pombo V, Barrios R, Pavani C. Photobiomodulation in the treatment of palmar-plantar erythrodysesthesia: a randomised controlled clinical study protocol. BMJ Open. 2024 Apr 23;14(4):e081459. doi: 10.1136/bmjopen-2023-081459. PMID 38657999